CLINICAL TRIAL: NCT06347549
Title: Diaphragmatic and Sternocleidomastoid Muscle Recruitment at Various Inspiratory Loads With and Without Breathing Instruction in Healthy Adults
Brief Title: The Impact of Diaphragmatic Breathing Instructions and Inspiratory Pressures on Diaphragm Contraction in Healthy Adults
Status: Completed | Type: Observational
Sponsor: Hong Kong Metropolitan University (Other)
Responsible Party: Principal Investigator, LIU FANG, PhD student, Hong Kong Metropolitan University
Other Study IDs: HE-SF2024/09
Record Dates: First submitted 2024-03-28; First posted 2024-04-04 (Actual); Last update posted 2025-01-28 (Actual); Status verified 2025-01

CONDITIONS: Diaphragm
Keywords: Diaphragmatic thickening fraction; Sternocleidomastoid muscles; Inspiratory pressures

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Healthy adults: Participants ≥18 years of age with normal health will be recruited in this study.
  Interventions: Diagnostic Test: Various intensities of inspiratory muscle training

INTERVENTIONS:
Diagnostic Test: Various intensities of inspiratory muscle training — Each participant will be instructed to use a pressure threshold inspiratory loading device to perform, in random order, 10 breaths at an inspiratory intensity of 30%, 40%, 50%, 60%, 70%, and 80% of their maximum inspiratory pressure (MIP). A rest period of 15 minutes will be allowed between each inspiratory pressure set of 10 breaths. Simultaneous surface electromyographic (sEMG) recording of the right sternocleidomastoid muscle and ultrasound of right diaphragmatic thickness will be conducted during each breath.
  The entire recording procedure will be repeated on a separate day. During the repeat measurements, participants will be provided with specific breathing instruction to focus on the use of the diaphragm and to inhale air to the lower part of the chest.

SUMMARY:
This is a cross-sectional obsessional study.

This study aims (1) to investigate the relationship between sternocleidomastoid muscle recruitment and diaphragm thickness fraction during increasing inspiratory resistance in healthy adults; (2) to compare diaphragmatic and sternocleidomastoid muscle recruitment patterns with and without a standard diaphragmatic breathing instruction with increasing inspiratory resistance in healthy adults.

Participants will be asked to breathe through a pressure threshold inspiratory loading device under different inspiratory resistances with and without a standard diaphragmatic breathing instruction. sternocleidomastoid muscle activity will be measured with surface electromyography, and diaphragm thickness will be assessed with ultrasonography.

DETAILED DESCRIPTION:
Upon arrival at the laboratory, eligible participants will first perform a standard spirometry lung function test. The maximum inspiratory pressure (MIP) will be determined with a pressure threshold inspiratory loading device (POWERbreathe, K2). Each participant will then be instructed to use the device to perform, in random order, 10 breaths at an inspiratory intensity of 30%, 40%, 50%, 60%, 70%, and 80% MIP. A rest period of 15 minutes will be allowed between each inspiratory pressure set of 10 breaths. Simultaneous surface electromyographic (sEMG) recording of the right sternocleidomastoid muscle and ultrasound of right diaphragmatic thickness will be conducted during each breath.

The entire recording procedure will be repeated on a separate day. During the repeat measurements, participants will be provided with specific breathing instruction to focus on the use of the diaphragm and to inhale air to the lower part of the chest. Practice trials will be conducted to ensure participant's understanding of diaphragmatic breathing.

ELIGIBILITY:
Inclusion Criteria:

* Participants ≥18 years of age with normal health

Exclusion Criteria:

* Pregnancy.
* Participants with known cardiovascular, pulmonary, musculoskeletal or psychiatric disorders.
* Participants with respiratory symptoms (from flu or other respiratory infection during the 2 weeks prior to measurements.
* Participants can not cooperate the maximal inspiratory pressure measurement.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy adults
Sampling Method: Probability Sample
Enrollment: 62 (Actual)
Dates: Start 2024-04-08 (Actual); Primary Completion 2024-07-16 (Actual); Study Completion 2024-07-16 (Actual)

PRIMARY OUTCOMES:
Diaphragmatic thickening fraction | Through study completion, an average of 1 year
  Diaphragmatic thickening fraction is determined by "(thickness of the diaphragm at end inspiratory - thickness at end expiratory)/thickness at end expiratory". Diaphragmatic thickness will be measured by ultrasonography.

SECONDARY OUTCOMES:
Muscle activation of the sternocleidomastoid muscle | Through study completion, an average of 1 year
  Surface electromyography will be used to measure accessory inspiratory muscle (sternocleidomastoid muscles) activity during each inspiratory muscle training intensity.
Perceived Exertion Borg scale | Through study completion, an average of 1 year
  This is a vertical scale quantified from 0 to 10, where 0 represents no symptoms, and 10 represents the maximum symptoms. The Borg score provides an individual measurement of the exercise intensity.

CONTACTS AND LOCATIONS:
Overall Officials: William Tsang, Principal Investigator — Hong Kong Metropolitan University
Locations (1):
- Hong Kong Metropolitan University, Hong Kong, None Selected, China

IPD SHARING:
Plan to Share IPD: Undecided

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-03-25): https://cdn.clinicaltrials.gov/large-docs/49/NCT06347549/Prot_SAP_000.pdf
  • Informed Consent Form (2024-03-25): https://cdn.clinicaltrials.gov/large-docs/49/NCT06347549/ICF_001.pdf